CLINICAL TRIAL: NCT03779516
Title: Effect of Preoperative Nebulized Lidocaine on Postoperative Sore Throat After Endotracheal Intubation
Brief Title: Effect of Nebulized Lidocaine on Postoperative Sore Throat
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in procedure
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AntalyaTRH 28
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2018-12

CONDITIONS: Sore Throat
MeSH Terms: conditions — Pharyngitis | interventions — Sodium Chloride; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group C (Active Comparator): In Control Group, 4 mL of saline solution was administered using a face mask and a compressed gas-powered jet nebulizer for 15 min
  Interventions: Other: Saline
- Group L (Active Comparator): In Lidocaine Group 4 mL of 4% lidocaine was administered using a face mask and a compressed gas-powered jet nebulizer for 15 min
  Interventions: Other: Lidocaine

INTERVENTIONS:
Other: Saline — Effect of saline on postoperative sore throat
  Arms: Group C
Other: Lidocaine — Effect of nebulized lidocaine on postoperative sore throat
  Arms: Group L

SUMMARY:
The purpose of this study is to test the hypothesis that use of preoperative nebulized lidocaine is reduced the incidence of postoperative sore throat after endotracheal intubation.

DETAILED DESCRIPTION:
Adult patients undergoing video-assisted thoracic surgery (VATS) requiring double lumen tube (DLT) endotracheal intubation for one-lung ventilation (OLV) were enrolled in the study. Patients were randomized by means of computer-generated order randomization into two groups: Group C (those who received a saline solution as placebo delivered by nebulization) and Group L (those who received lidocaine delivered by nebulization).

At 1, 6 and 24 h after tracheal extubation, an observer blinded to treatments evaluated the patients in terms of sore throat and hoarseness. In addition, Patients' satisfaction, intraoperative and postoperative opioid and analgesics consumption and complaints such as dysphagia, nausea and vomiting were recorded. Hemodynamic variables such as blood pressure and heart rate were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing video-assisted thoracic surgery requiring double lumen tube endotracheal intubation for one-lung ventilation
* American Society of Anesthesiologists class 1,2 and 3
* Ability to consent

Exclusion Criteria:

* patients <18 years old
* body mass index (BMI) <20 or >35 kg/m2
* Mallampati grade 3 or 4
* mouth opening < 3 cm
* preexisting hoarseness or sore throat
* coagulopathy
* patient with upper respiratory tract infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Changes in the incidence of postoperative sore throat | 24 hours
  Sore throat was assessed using a 0-100 mm visual analog scale (VAS), where a score of 0 represents no pain and a score of 100 reflects the worst pain imaginable.

SECONDARY OUTCOMES:
whether the hoarseness was present or not | 24 hours
  Hoarseness was defined as a change in voice quality and it was assessed by the patients themselves. The change in voice quality at any time during the observation period was defined as "hoarseness was present".
Intraoperative opioid consumption | 60 minutes
  Assessed in intraoperative period
Postoperative analgesic consumption | 24 hours
  Assessed in postoperative period
Changes in mean arterial pressure | 60 minutes
  Assessed every 5 minutes during the procedure
Changes in heart rate | 60 minutes
  Assessed every 5 minutes during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sait Kavakli, MD, Principal Investigator — Antalya Training and Research Hospital; Hilal Yavuzel, MD, Principal Investigator — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital; Ulku Arslan, MD, Principal Investigator — Karabuk University Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)